CLINICAL TRIAL: NCT06837155
Title: A QT/QTc Evaluation Study of TS-172 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TS172-03-07
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TS-172 20 mg (Experimental)
  Interventions: Drug: TS-172 20 mg
- TS-172 90 mg (Experimental)
  Interventions: Drug: TS-172 90 mg
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-172 20 mg — oral administration of TS-172 20 mg
  Arms: TS-172 20 mg
Drug: TS-172 90 mg — oral administration of TS-172 90 mg
  Arms: TS-172 90 mg
Drug: Moxifloxacin — oral administration of moxifloxacin 400 mg
  Arms: Moxifloxacin
Drug: Placebo — oral administration of placebo
  Arms: Placebo

SUMMARY:
A clinical study to evaluate the effects on QT/QTc interval of TS-172 in healthy adults subjects

ELIGIBILITY:
Inclusion criteria

1. Japanese healthy subjects aged =>18 and <40 years at the time of obtaining informed consent
2. Subjects whose body weight is >=40 kg at the screening test, and body mass index is >=18.5 and <25.0
3. Subjects with both heart rates are =>45 and =<100 beats/min on a standard 12-lead electrocardiogram at the screening test and before drug administration in Period 1

Exclusion criteria

1. Subjects with a history of hypersensitivity to moxifloxacin or other quinolone antibiotics
2. Subjects with a family history or risk factors for aortic aneurysm or aortic dissection (e.g., Marfan syndrome)
3. Subjects with a family history of sudden death
4. Subjects with congenital diseases, heart diseases, or medical history of such conditions
5. Subjects with risk factors for Torsades de Pointes (TdP) (e.g., heart failure, hypokalemia, or a family history of long QT syndrome) or medical history of such conditions
6. Subjects with medical history of syncope suspected to be related to TdP, unexplained syncope, or seizures
7. Subjects with standard 12-lead electrocardiogram waveforms that make it difficult to evaluate QTc prolongation (e.g., drift, EMG interference, T wave morphology, significant sinus arrhythmia, or frequent ectopic beats) at the screening and before the administration of the study drug in Period 1
8. Subjects with a QTcF (QT interval corrected using Fridericia's formula) of =>450 msec in the standard 12-lead ECG test at the screening and before the administration of the study drug in Period 1

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
QTcF:QT-interval corrected by Fridericia corrections in Holter ECGs | Up to 24 hours postdose during each period

CONTACTS AND LOCATIONS:
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No